CLINICAL TRIAL: NCT06538181
Title: A Phase 1 Study of Pacritinib in Vacuoles, E1 Ubiqutin-activating Enzyme, X-linked, Autoinflammatory, Somatic (VEXAS) Syndrome
Brief Title: Pacritinib in Vacuoles, E1 Ubiqutin-activating Enzyme, X-linked, Autoinflammatory, Somatic (VEXAS) Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202412141
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: E1 Ubiqutin-activating Enzyme, X-linked, Autoinflammatory, Somatic Syndrome; VEXAS; Vexas Syndrome
Keywords: VEXAS; Autoinflammatory; UBA1; Pacritinib
MeSH Terms: conditions — VEXAS syndrome | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose De-Escalation (Safety Run-in): Pacritinib (Experimental): Assigned dose of pacritinib by mouth twice per day. Each cycle is 28 days and participants can receive up to 12 cycles of treatment.
- Dose Expansion: Pacritinib (Experimental): Recommended phase II dose of pacritinib by mouth twice per day. Each cycle is 28 days and participants can receive up to 12 cycles of treatment.

INTERVENTIONS:
Drug: Pacritinib — Starting dose is 200 mg twice per day by mouth. Dose level -1 is 100 mg twice per day by mouth.

SUMMARY:
VEXAS (vacuoles, E1 ubiqutin-activating enzyme, X-linked, autoinflammatory, somatic syndrome) is a recently described disorder with severe hematologic and rheumatologic manifestations caused by somatic variants in the ubiquitin- activating enzyme gene, UBA1, that is acquired in hematopoietic progenitor cells. Patients are often debilitated by autoinflammatory symptoms and there is currently no standard of care available. There is a clinically unmet need for better therapies in VEXAS Syndrome. There have been no prospective clinical trials of JAK-I in VEXAS syndrome. The investigators hypothesize that pacritinib, as a JAK2/IRAK1 inhibitor with a manageable safety profile in myelofibrosis patients with thrombocytopenia, will improve the autoinflammatory and hematologic manifestations of VEXAS syndrome with a tolerable toxicity profile.

The investigators propose a single arm, pilot Phase 1 study evaluating the safety and tolerability of pacritinib in patients with VEXAS syndrome with an initial safety run-in phase of 6 patients treated with pacritinib 200mg twice daily (BID) on days 1-28 of a continuous 28 day cycle. If no more than 1 patient experiences a dose-limiting toxicity (DLT), the investigators will enroll an expansion cohort to gain additional toxicity and efficacy data, for a total enrollment of 15 patients. If more than 1 patient experiences a DLT during the safety run-in phase, the investigators will decrease the dose to 100 mg BID, and if no more than 1 of 6 patients experiences a DLT, the investigators will complete the expansion cohort as above for up to a total enrollment of 15 patients. If more than 1 patient experiences a DLT at 100 mg BID, the investigators will discontinue the study. Patients will be treated for up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have UBA1 mutation with a variant allele frequency (VAF) of ≥ 2% detected on a next generation sequencing panel and have at least one of the following current or past clinical manifestation of VEXAS syndrome, as determined by the attending physician:

  * skin rash
  * vasculitis
  * chondritis
  * ocular/orbital inflammation (e.g., uveitis/iritis, episcleritis)
  * genitourinary inflammation (e.g., epididymitis/orchitis)
  * arthritis/arthralgias
  * pulmonary inflammation (e.g., alveolitis/pleural effusion,)
  * fever
  * thrombosis
  * splenomegaly
  * hepatomegaly
  * myocarditis or pericarditis
  * cytopenias (defined as hemoglobin <11 g/dL, platelets < 100 X 10^9 /L, OR absolute neutrophil count <1.0 X 10^9 /L).
* Patients with VEXAS syndrome who have never been treated with a JAK-I will be eligible to enroll on study. A stable corticosteroid dose must be maintained for at least 14 days prior to start of pacritinib.
* Patients who have previously been treated with a JAK-I other than pacritinib, or who are currently being treated with a JAK-I other than pacritinib, may be eligible after a 28 day washout if either (i) their symptoms are not adequately controlled, as determined by the treating physician, or (ii) they have been unable to taper corticosteroids to an equivalent of <10 mg prednisone/day, and in the opinion of the treating physician, may benefit from a change in JAK-I. A stable corticosteroid dose must be maintained for at least 14 days prior to start of pacritinib.
* At least 18 years of age.
* ECOG performance status ≤ 3.
* Organ function as defined below:

  * Absolute neutrophil count ≥ 0.5 K/cumm
  * Platelets ≥ 25 K/cumm
  * PT/PTT <2.5 X upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
* QTcF < 480 msec.
* The effects of pacritinib on the developing human fetus are unknown. For this reason and because pacritinib was shown to be teratogenic in animal studies, women of childbearing potential and men must agree to use highly effective contraception prior to study entry, for the duration of study participation, and for 30 days after completion of study treatment. Hormonal contraception is no longer considered highly effective alone as pacritinib is a CYP3A4 inducer and accelerated progesterone metabolism. The contraceptive methods considered highly effective for WOCBP who receive pacritinib are intrauterine devices, bilateral tubal occlusion, vasectomized partner, or total sexual abstinence. Hormonal contraceptives (e.g., Depo-Provera) alone are not considered highly effective methods of contraception on their own when in treatment with pacritinib; such hormonal contraceptives must be combined with an additional barrier method (condom, diaphragm with spermicidal gel, or condoms with spermicides to be considered highly effective. Highly effective contraceptive methods in males include vasectomy, sexual abstinence, and condoms when combined with their partner using a highly effective method (including oral contraceptives).
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document or that of legally authorized representative, if applicable.
* Patients with myelodysplastic neoplasms (MDS) or plasma cell dyscrasias are eligible if they are not undergoing active treatment. Supportive care is permitted.

Exclusion Criteria:

* Prior use of pacritinib.
* Use of another JAK inhibitor within 28 days of C1D1 of pacritinib.
* Currently receiving any other investigational agents. Patients may be eligible after 28 day washout.
* Thrombotic events (arterial or venous) within 60 days prior to enrollment.
* Any recent clinically significant bleeding within at least 7 days prior to enrollment.
* Any active or acute infection.
* History of malignancy within the prior 2 years, with the exception of MDS and plasma cell dyscrasias, or non-melanoma skin cancers that have been treated.
* History of clinically significant cardiovascular disease or clinically significant abnormalities in rhythm or conduction during screening EKG, including severe cardiac events, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or heart failure.
* Currently receiving immunosuppressants (other than corticosteroids), disease-modifying antirheumatic drugs (DMARDs), or biologic cytokine inhibitors. Patients may be eligible after 28 day washout.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pacritinib.
* Concurrent use of strong CYP3A4 inhibitors or inducers. Patients may be eligible after washout period of 28 days (or 5 half-lives, whichever is shorter).
* Diagnosis or history of moderate (Child-Pugh B) and severe hepatic impairment (Child-Pugh C).
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of C1D1 or negative urine pregnancy test within 3 days of C1D1.
* Known active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Patients with latent tuberculosis. Patients must have a negative T-Spot during screening to be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | Through completion of cycle 1 (estimated to be 28 days)
  Dose-limiting toxicities (DLTs) are adverse events defined by the protocol that occur during the DLT observation period (Cycle 1) of the study, unless clearly attributable to underlying disease or another cause unrelated to the study.
Recommended phase II dose (RP2D) | Through completion of cycle 1 (each cycle is 28 days) for all treated participants
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity (DLT) during the first cycle. The recommended phase II dose (RP2D) will be less than or equal to the MTD. If the MTD is not reached, and in the opinion of the investigators, the toxicity profile is acceptable, Dose Level 1 will be the RP2D.

SECONDARY OUTCOMES:
Change in white blood cell count | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in absolute neutrophil count | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in absolute lymphocyte count | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in hemoglobin | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in platelets | Baseline, 1 month, 3 months, 6 months, and 12 months
Number of participants with hematologic improvement as measured with neutrophils | Through completion of treatment (estimated to be 12 months)
  Using IWG 2018 criteria
Number of participants with hematologic improvement as measured with hemoglobin | Through completion of treatment (estimated to be 12 months)
  Using IWG 2018 criteria
Number of participants with hematologic improvement as measured with platelets | Through completion of treatment (estimated to be 12 months)
  Using IWG 2018 criteria
UBA1 variant allele frequency | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in C reactive protein (CRP) | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in ferritin | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in ESR | Baseline, 1 month, 3 months, 6 months, and 12 months
Change in inflammatory and rheumatologic symptoms as measured by the VEXAS Disease Activity Index | Baseline, 1 month, 3 months, 6 months, and 12 months
Time to next treatment | Through completion of follow-up (estimated to be 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Meagan A Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Data 9 available months to 36 months after publication
Access Criteria: Investigators who proposed use of the data has been approved by independent review committee identified for this purpose

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu